CLINICAL TRIAL: NCT02036957
Title: EFFECTIVENESS OF MARY D'UOL REPAIR BALM FOR PREVENTING AND / OR REDUCING TOXICITY SKIN IN PATIENTS WITH CANCER AND TREATMENT WITH ANY Antineoplastic Agent. RANDOM CLINICAL TRIAL.
Brief Title: MARY DUOL REPAIR BALM IN THE PREVENTION OR REDUCING ANTINEOPLASIC AGENTS' SKIN TOXICITY
Acronym: B-DUOL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Patricia Seoane, oncologist physician, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-01
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Dermatitis, Adverse Drug Reaction
Keywords: capecitabine; dermatologic toxicity
MeSH Terms: conditions — Drug Eruptions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BALM ARM (Experimental): The product will be applied throughout the body in abundant quantity to achieve that the skin be perfectly hydrated. Will be applied twice a day (after showering and at night), massaging the area until completely absorption.
  Interventions: Procedure: BALM ARM
- PLACEBO ARM (Placebo Comparator): It be applicated in like manner that balm arm
  Interventions: Procedure: PLACEBO ARM

INTERVENTIONS:
Procedure: BALM ARM — The product will be applied throughout the body in abundant quantity to achieve that the skin be perfectly hydrated. The product will be applied twice a day (after showering in the morning and at night), massaging the area until completely absorption. Treatment will last three months, and at this time, We will measure toxicologic toxicity in both arms.
  Arms: BALM ARM
Procedure: PLACEBO ARM — The product will be applied throughout the body in abundant quantity to achieve that the skin be perfectly hydrated. The product will be applied twice a day (after showering in the morning and at night), massaging the area until completely absorption. Treatment will last three months, and at this time, We will measure toxicologic toxicity in both arms.
  Arms: PLACEBO ARM

SUMMARY:
Capecitabine is a drug that produces dermatologic toxicity frequently (palmoplantar erythrodysesthesia, rash , alopecia , erythema , dryness, pruritus, hyperpigmentation , rash, peeling , dermatitis , abnormal pigmentation, and less often blistering, skin ulcers , photosensitivity reactions, swelling of the face and purple) . The impact in patients' quality of life is great, so We had decided to conduct a randomized clinical trial to evaluate the effectiveness Mary D' uol balm preventing dermatologic toxicity in patient treated with capecitabine .

Design: Randomized clinical trial phase II, in parallel and double-blind groups

Target population : Patients with colon cancer stage II or III ( Dukes' C ) , who will initiate treatment with capecitabine monotherapy.

Inclusion criteria: Over 18 years, II or III colon (Dukes' C) colon cancer, primary diagnosis, capecitabine monotherapy, sign the informed consent.

Primary endpoint: Dermatologic toxicity (yes / no) Statistical analysis: The primary endpoint (percentage of patients that develop dermalogic toxocity in both groups) will be analyzed by a logistics regression model

DETAILED DESCRIPTION:
Intervention: Preventive treatment of dermatologic toxicities begin on the day of initiation of treatment with Xeloda, capecitabine + oxaliplatin, Adriamycin Liposomial or cytarabine

The product will be applied throughout the body in abundant quantities so that the skin is perfectly hydrated. It is applied twice daily (after showering and evening), gently massaging the area until completely absorbed.

The product will be provided at the unit of oncology pharmacy, when the patient is randomized. 3 packs per cycle will be provided. If not enough (because the patient has greater surface area) will be supplied more. Each time you start a new cycle 3 new packages will be delivered.

The patient will not apply any other cosmetic product in the treated areas.

In addition all patients regardless of the group will receive recommendations for reducing the appearance of skin problems caused by these type of drugs.

The study will have a total duration of 24 weeks (8 cycles of chemotherapy), except in cases of patients requiring a cycle delay for filing toxicity. In these patients the total duration of the study must be sufficient to end the eighth cycle.

If the side effects are so severe that greatly affect the quality of life of the patient and the doctor thinks fit, may prescribe drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* Sign the informed consent

Exclusion Criteria:

* Patients with neoadjuvant treatment.
* Patients with dermatologic diseases.
* Patients treated with corticosteroids.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who develop dermatologic toxicity. | 3 moths
  Compare the percentage of patients who develop dermatologic toxicity in any grade (1-5) between intervention and control group at three months of starting treatment, through CTCAE scale (National Cancer Institute Common Toxicity Criteria).

SECONDARY OUTCOMES:
Need of pharmacological treatment to mitigate toxicity | 3 months
  Compare the percentage of patients in both groups who required pharmacological treatment to mitigate the dermatologic toxicity produced by chemotherapy
Quality of life | 3 months
  Compare the quality of life in both groups at three months, through the Skindex 29 scale to evaluate the quality of life due to skin disease.
Percentaje of patients who have reduces skin toxicity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Arantza Sáez de la Fuente, Msc, Study Chair — Basque Health Service (Research Unit); Patricia Seaone, MD, Principal Investigator — Basque Health Service (Research Unit); Raquel Cobos, Msc, Study Chair — Basque Health Service (Research Unit)
Locations (1):
- University hospital of Araba, Vitoria-Gasteiz, Álava, Spain